CLINICAL TRIAL: NCT00867490
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of a 4 Week Therapy With Aliskiren 300 mg Plus Hydrochlorothiazide 25 mg in Hypertensive Patients Not Adequately Responding to a 4 Week Therapy With Candesartan 32 mg Plus Hydrochlorothiazide 25 mg
Brief Title: Safety and Efficacy of Aliskiren + Hydrochlorothiazide (± Amlodipine 5 mg) in Patients With Moderate Hypertension
Acronym: AMAZING
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPH100ADE01
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2011-02-01 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Hypertension; aliskiren; cardiovascular diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

ARMS (1):
- Candesartan+HCTZ, aliskiren+HCTZ, aliskiren+HCTZ+amlodipine (Experimental)
  Interventions: Drug: Candesartan+HCTZ - Phase 1; Drug: Aliskiren+HCTZ - Phase 2; Drug: Aliskiren+HCTZ+amlodipine - Phase 3

INTERVENTIONS:
Drug: Candesartan+HCTZ - Phase 1 — 4 weeks treatment with candesartan 32 mg (two 16 mg tablets) plus hydrochlorothiazide 25 mg (two 12.5 mg tablets) taken orally with water in the morning between 7 and 10 am.
Drug: Aliskiren+HCTZ - Phase 2 — Patients with uncontrolled mean sitting diastolic blood pressure (msDBP ≥ 90 mm Hg) at the end of Phase 1 were treated for 4 weeks with aliskiren 300 mg plus hydrochlorothiazide 25 mg in a single tablet taken orally with water in the morning between 7 and 10 am.
Drug: Aliskiren+HCTZ+amlodipine - Phase 3 — The first 60 patients with uncontrolled mean sitting systolic or diastolic blood pressure (msDBP ≥ 90 mm Hg and/or msSBP ≥ 140 mm Hg) at the end of Phase 2 were offered 4 weeks treatment with aliskiren 300 mg plus HCTZ 25 mg in a single tablet plus an amlodipine 5 mg tablet taken orally with water in the morning between 7 and 10 am.

SUMMARY:
This study will assess the safety and efficacy of aliskiren plus hydrochlorothiazide (HCTZ) in patients who do not achieve controlled blood pressure levels after treatment with another specified antihypertensive medication. There was an optional study extension for the first eligible 60 patients who wanted to participate that contains the triple therapy with amlodipine 5 mg and aliskiren 300 mg plus HCTZ 25 mg.

DETAILED DESCRIPTION:
Title of study extension: An open-label, multicenter extension to evaluate the efficacy and safety of a 4 week therapy with amlodipine 5 mg and aliskiren 300 mg plus HCTZ 25 mg in hypertensive patients not adequately responding to a 4 week therapy each with the combinations of candesartan 32 mg plus hydrochlorothiazide 25 mg followed by aliskiren 300mg plus hydrochlorothiazide 25 mg

ELIGIBILITY:
Inclusion Criteria for Core Study:

- Patients with mean sitting diastolic blood pressure ≥ 100 mmHg and < 110 mmHg

Inclusion criteria for the Extension:

- msSBP ≥ 140 mm Hg and/or msDBP ≥ 90 mm Hg at Visit 5 of the core study

Exclusion Criteria for Core Study:

* Patients with mean diastolic blood pressure ≥ 110 mmHg or mean systolic blood pressure ≥ 180 mmHg
* Patients with prior stroke, hypertensive encephalopathy or heart attack
* Patients with type 1 diabetes mellitus
* Patients with type 2 diabetes mellitus with poor glucose control

Exclusion criteria for the Extension:

* Premature discontinuation in the core study or failure to comply with the core study protocol
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures, known or suspected contraindications to diuretics as described in the SmPC (particularly amlodipine 5 mg), e.g. severe hypotension, shock - including cardiogenic shock, obstructions impairing the flow out of the left ventricle (e.g. significant aortic stenosis)
* Any patient that the investigator decides should not participate in the extension study for medical reasons

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Investigative Site, Chemnitz, Germany

REFERENCES:
- [Derived] Schweizer J, Ulmer HJ, Benduhn H, Klebs S. Efficacy and tolerability of aliskiren 300 mg/hydrochlorothiazide 25 mg (+/- amlodipine 5 mg) in hypertensive patients not controlled by candesartan 32 mg plus HCT 25 mg. Curr Med Res Opin. 2011 Jan;27(1):131-40. doi: 10.1185/03007995.2010.537318. Epub 2010 Nov 30. PMID 21117946

RESULTS

PARTICIPANT FLOW:
Groups:
- Candesartan+HCTZ, Aliskiren+HCTZ, Aliskiren+HCTZ+Amlodipine: 4 weeks treatment with candesartan 32 mg plus hydrochlorothiazide (HCTZ) 25 mg (Phase 1) followed by 4 weeks treatment with aliskiren 300 mg plus HCTZ 25 mg (Phase 2) in patients with uncontrolled diastolic blood pressure (BP) in Phase 1 followed by (optional) 4 weeks treatment with aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg (Phase 3) in patients with uncontrolled systolic or diastolic BP in Phase 2.
Period: Phase 1 - Candesartan+HCTZ
Arm/Group | Candesartan+HCTZ, Aliskiren+HCTZ, Aliskiren+HCTZ+Amlodipine
Started | 186
Completed | 176
Not Completed | 10
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 4
Not completed — Administrative Problems | 1
Period: Phase 2 - Aliskiren+HCTZ
Arm/Group | Candesartan+HCTZ, Aliskiren+HCTZ, Aliskiren+HCTZ+Amlodipine
Started | 123 (Only patients with mean sitting diastolic BP ≥ 90 mmHg at the end of Phase 1 entered this phase.)
Completed | 120
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Phase 3 - Aliskiren+HCTZ+Amlodipine
Arm/Group | Candesartan+HCTZ, Aliskiren+HCTZ, Aliskiren+HCTZ+Amlodipine
Started | 61 (The first 60 patients with systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg entered this phase.)
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Candesartan+HCTZ, Aliskiren+HCTZ, Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 186
Age Continuous [Mean (Standard Deviation); unit: years]
  Phase I - Candesartan+HCTZ | 56.2 (10.62)
  Phase II - Aliskiren+HCTZ | 57.4 (10.87)
  Phase III - Aliskiren+HCTZ+amlodipine | 58.9 (10.31)
Sex/Gender, Customized [Number; unit: Participants] — Female
  Participants
    Phase I - Candesartan+HCTZ | 78
    Phase II - Aliskiren+HCTZ | 48
    Phase III - Aliskiren+HCTZ+amlodipine | 24
Sex/Gender, Customized [Number; unit: Participants] — Male
  Participants
    Phase I - Candesartan+HCTZ | 108
    Phase II - Aliskiren+HCTZ | 75
    Phase III - Aliskiren+HCTZ+amlodipine | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) During the Core Phase of the Study
Description: The arm in which the highest sitting diastolic pressures were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, systolic/diastolic blood pressure were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements. A negative change indicates improvement.
Time Frame: Baseline Phase 2 to end of Phase 2
Population: Intent-to-treat population (ITT): All patients who took at least one dose of aliskiren plus HCTZ who had at least one primary efficacy parameter evaluation. Patients who dropped out were included in the ITT population if there was any BP measurement available; their last available blood pressure measurement was used for the analysis.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Phase 2 - Aliskiren+HCTZ: Patients with uncontrolled mean sitting diastolic BP (msDBP ≥ 90 mm Hg) at the end of Phase 1 were treated for 4 weeks with aliskiren 300 mg plus hydrochlorothiazide (HCTZ) 25 mg in a single tablet taken orally with water in the morning between 7 and 10 am.
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
mmHg | -3.12 [-4.29 to -1.95]

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) During the Core Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 2 to end of Phase 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
mmHg | -2.81 [-4.81 to -0.81]

3. Secondary Outcome: Change in Sitting Pulse Pressure During the Core Phase of the Study
Description: Pulse pressure is systolic pressure (SP) minus diastolic pressure (DP). The arm in which the highest sitting DPs were found at study entry was the arm used for all subsequent readings. A calibrated sphygmomanometer and appropriate size cuff were used to measure arterial sitting blood pressure (BP) at trough with the arm supported at the level of the heart. At each study visit, after having the patient in a sitting position for at least 5 minutes, SP and DP were measured 3 times at 1-2 minute intervals. A mean was calculated from the 3 measurements. A negative change indicates improvement.
Time Frame: Baseline Phase 2 to end of Phase 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
mmHg | 0.31 [-1.39 to 2.01]

4. Secondary Outcome: Change in Sitting Pulse Rate During the Core Phase of the Study
Description: Pulse rate was measured once for 30 seconds just prior to blood pressure measurements in the sitting position.
Time Frame: Baseline Phase 2 to end of Phase 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: BPM (beats per minute)
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
BPM (beats per minute) | 0.27 [-1.15 to 1.69]

5. Secondary Outcome: Percentage of Patients Who Achieved Normalized Blood Pressure During the Core Phase of the Study
Description: Normalized blood pressure was defined as a msSBP < 140 mmHg and/or a msDBP < 90 mmHg.
Time Frame: Baseline Phase 2 to end of Phase 2
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
Percentage of patients
  msSBP < 140 mmHg | 37.4
  msDBP < 90 mmHg | 33.3

6. Secondary Outcome: Percentage of Patients Who Achieved a Protocol-defined Blood Pressure Response During the Core Phase of the Study
Description: Blood pressure response was defined as msSBP < 140 mmHg or a 20 mmHg decrease in msSBP at the end of Phase 2 compared to Baseline in Phase 2 or a msDBP < 90 mmHg or a 10 mmHg decrease in msDBP at the end of Phase 2 compared to Baseline in Phase 2.
Time Frame: Baseline Phase 2 to end of Phase 2
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Phase 2 - Aliskiren+HCTZ
Number analyzed (Participants) | 123
Percentage of patients
  msSBP response | 37.4
  msDBP response | 34.1

7. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) During the Extension Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Phase III - Aliskiren+HCTZ+Amlodipine: The first 60 patients with uncontrolled mean sitting systolic or diastolic blood pressure (msDBP ≥ 90 mm Hg and/or msSBP ≥ 140 mm Hg) at the end of Phase 2 were offered a 4 week treatment extension with aliskiren 300 mg plus hydrochlorothiazide (HCTZ) 25 mg in a single tablet plus amlodipine 5 mg tablet.
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
mmHg | -5.87 [-7.48 to -4.26]

8. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) During the Extension Phase of the Study
Description: as for outcome 1
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
mmHg | -9.20 [-11.86 to -6.54]

9. Secondary Outcome: Change in Sitting Pulse Pressure During the Extension Phase of the Study
Description: as for outcome 3
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
mmHg | -3.33 [-5.40 to -1.27]

10. Secondary Outcome: Change in Sitting Pulse Rate During the Extension Phase of the Study
Description: Pulse rate was measured once for 30 seconds just prior to blood pressure measurements in the sitting position.
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Mean (95% Confidence Interval); unit: BPM (beats per minute)
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
BPM (beats per minute) | 0.03 [-1.82 to 1.89]

11. Secondary Outcome: Percentage of Patients Who Achieved Normalized Blood Pressure During the Core Phase of the Study
Description: Normalized was defined as a msSBP < 140 mm Hg and/or a msDBP < 90 mm Hg.
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Number; unit: Percentage of patients
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
Percentage of patients
  msSBP < 140 mmHg | 54.1
  msDBP < 90 mmHg | 44.3

12. Secondary Outcome: Percentage of Patients Who Achieved a Protocol-defined Blood Pressure Response During the Core Phase of the Study
Description: as for outcome 6
Time Frame: Baseline Phase 3 to end of Phase 3
Population: Safety population: All patients who took at least one dose of aliskiren 300 mg plus HCTZ 25 mg plus amlodipine 5 mg.
Measure: Number; unit: Percentage of patients
Arm/Group | Phase III - Aliskiren+HCTZ+Amlodipine
Number analyzed (Participants) | 61
Percentage of patients
  msSBP response | 54.1
  msDBP response | 47.5

ADVERSE EVENTS:
Groups:
- Phase 1 - Candesartan+HCTZ: 4 weeks treatment with candesartan 32 mg (two 16 mg tablets) plus hydrochlorothiazide (HCTZ) 25 mg (two 12.5 mg tablets) taken orally with water in the morning between 7 and 10 am.
- Phase 3 - Aliskiren+HCTZ+Amlodipine: The first 60 patients with uncontrolled mean sitting systolic or diastolic blood pressure (msDBP ≥ 90 mm Hg and/or msSBP ≥ 140 mm Hg) at the end of Phase 2 were offered a 4 week treatment extension with aliskiren 300 mg plus hydrochlorothiazide (HCTZ) 25 mg in a single tablet plus amlodipine 5 mg tablet taken orally with water in the morning between 7 and 10 am.
Arm/Group | Phase 1 - Candesartan+HCTZ | Phase 2 - Aliskiren+HCTZ | Phase 3 - Aliskiren+HCTZ+Amlodipine
Serious Adverse Events (participants affected / at risk) | 1/186 | 2/123 | 0/61
Other Adverse Events (participants affected / at risk) | 0/186 | 0/123 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - Candesartan+HCTZ (N=186) | Phase 2 - Aliskiren+HCTZ (N=123) | Phase 3 - Aliskiren+HCTZ+Amlodipine (N=61)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The Phases of this study were entered in separate tables for outcomes and the Phases for SAEs and the AEs were entered all in one table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.